CLINICAL TRIAL: NCT05706103
Title: Efficacy of Specific Skilled Motor Versus General Exercise Training on Peripheral Muscle and Central Brain Alterations in Patients with Recurrent Low Back Pain
Brief Title: Exercise Therapy for Recurrent Low Back Pain: Unraveling the Puzzle of Peripheral Muscle and Central Brain Changes (B670201420984)
Acronym: ExTraS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Fund for Scientific Research, Flanders, Belgium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BC-05152; U1111-1283-4631 (Registry Identifier: Universal Trial Number (UTN))
Record Dates: First submitted 2021-11-24; First posted 2023-01-31 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Low Back Pain, Recurrent
Keywords: low back pain; motor control; exercise; randomized controlled trial
MeSH Terms: conditions — Low Back Pain; Motor Activity

STUDY DESIGN:
Intervention Model Description: The study model is parallel. Participants experiencing recurrent LBP patients will be randomly allocated (1:1) to receive either specific skilled motor training or general extension training (i.e. parallel study model). Both groups will first receive low-load training (i.e. at 25-30% of the individual's repetition maximum, sessions 1-9) followed by high-load training (i.e. at 40-60% of the individual's one repetition maximum, sessions 10-18) (i.e. cross-over study model).
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Specific skilled motor training (Experimental): 13 weeks of treatment, with 18 supervised treatment sessions in combination with an individualized home-exercise program. This group will first receive low-load training (i.e. at 25-30% of the individual's repetition maximum, sessions 1-9) followed by high-load training (i.e. at 40-60% of the individual's one repetition maximum, sessions 10-18).
  Interventions: Behavioral: Specific skilled motor training
- General extension training (Active Comparator): 13 weeks of treatment, with 18 supervised treatment sessions in combination with an individualized home-exercise program. This group will first receive low-load training (i.e. at 25-30% of the individual's repetition maximum, sessions 1-9) followed by high-load training (i.e. at 40-60% of the individual's one repetition maximum, sessions 10-18).
  Interventions: Behavioral: General extension training

INTERVENTIONS:
Behavioral: Specific skilled motor training — Participants allocated to the skilled motor training group will receive sensorimotor training of the intrinsic muscles of the lumbopelvic region, namely the multifidus, transversus abdominis, and pelvic floor muscles.
  Arms: Specific skilled motor training
Behavioral: General extension training — Participants allocated to the general extension training group will receive general training exercises using the David Back equipment from the Back Unit at Ghent University Hospital
  Arms: General extension training

SUMMARY:
Exercise therapy has been shown to be effective in decreasing pain and improving function for patients with recurrent low back pain (LBP). Research on the mechanisms that trigger and/or underlie the effects of exercise therapy on LBP problems is of critical importance for the prevention of recurring or persistence of this costly and common condition. One factor that seems to be crucial within this context is the dysfunction of the back muscles. Recent pioneering results have shown that individuals with recurring episodes of LBP have specific dysfunctions of these muscles (peripheral changes) and also dysfunctions at the cortical level (central changes). This work provides the foundation to take a fresh look at the interplay between peripheral and central aspects, and its potential involvement in exercise therapy. The current project will draw on this opportunity to address the following research questions: What are the immediate (after a single session) and the long-term effects (after 18 repeated sessions) of exercise training on: (1) back muscle structure; (2) back muscle function; (3) the structure of the brain; (4) and functional connectivity of the brain. This research project also aims to examine whether the effects are dependent on how the training was performed. Therefore a specific versus a general exercise program will be compared.

DETAILED DESCRIPTION:
Although the cause of persistent non-specific LBP remains unknown, structural and functional alterations of the brain and paravertebral muscles have been proposed as underlying mechanisms. As it is hypothesized that these alterations contribute to, or maintain non-specific LBP, exercise therapy is a key element in the rehabilitation of reoccurring LBP. Specific training of sensorimotor control of the lumbopelvic region (i.e. specific skilled motor training) has shown to decrease pain and disability in patients with LBP, but has not been found superior to other forms of exercise training regarding improvements in clinical outcome measures. On the other hand, this type of training seems to differentially impact the recruitment of the back muscles compared to general exercise training. However, research using multiple treatment sessions and including follow-up outcome assessments is scarce. Furthermore, it is unknown if improvements may be attributed to measurable peripheral changes in the muscle and/or central neural adaptations in the brain. The primary aim of this study is to examine the short and long-term effects of specific skilled motor control training versus unspecific general extension training on pain, functional disability, brain structure/function and muscle structure/function in recurrent LBP patients.

Method: In this double-blind, randomized controlled clinical trial 62 recurrent LBP patients will be randomly allocated (1:1) to receive either specific skilled motor training (i.e. the experimental group) or general extension training (i.e. control group). Each training group will receive 13 weeks of treatment, during which a total of 18 supervised treatment sessions will be delivered in combination with an individualized home-exercise program. Both groups will first receive low-load training (i.e. at 25-30% of the individual's repetition maximum, sessions 1-9) followed by high-load training (i.e. at 40-60% of the individual's one repetition maximum, sessions 10-18). Primary outcome measures include: LBP-related pain and disability (RMDQ, NRS and Margolis pain diagram), lumbar muscle structure and function (Dixon MRI and mf-MRI) and brain structure and function (MRI, DTI and fMRI). Secondary measures include: lumbopelvic control and proprioception (thoracolumbar dissociation test and position-reposition test), trunk muscle activity (RAM and QFRT) and psychosocial factors, including measures of physical activity (IPAQ-LF, SF-36), pain cognitions and perceptions (PCS, PCI and PVAQ), anxiety and depression (HADS), and kinesiophobia (TSK). Experimental data collection will be performed at baseline, immediately following the low-load training (i.e. after the 9th supervised treatment session), following the high-load training (i.e. after the 18th supervised treatment session), and at 3 months follow-up. Experimental data collection will comprise of magnetic resonance imaging of the brain and trunk muscles, clinical assessments assessing muscle function, and a battery of questionnaires evaluating psychosocial factors.

ELIGIBILITY:
Inclusion Criteria:

* History of non-specific recurrent LBP with the first onset being at least 6 months ago
* At least 2 episodes of LBP/year, with an 'episode' implying pain lasting a minimum of 24 hours which is preceded and followed by at least 1 month without LBP
* Minimum LBP intensity during episodes should be ≥2/10 on a numeric rating scale (NRS) from 0 to 10
* During remission the NRS intensity for LBP should be 0.
* LBP should be of that severity that it limits activities of daily living
* LBP should be of that severity that a (para)medic has been consulted at least once regarding the complaints
* Flexion pattern of LBP

Exclusion Criteria:

* Chronic LBP (i.e. duration remission <1 month)
* Subacute LBP (i.e. first onset between 3 and 6 months ago)
* Acute (i.e. first onset <3 months ago) LBP
* Specific LBP (i.e. LBP proportionate to an identifiable pathology, e.g. lumbar radiculopathy)
* Patients with neuropathic pain
* Patients with chronic widespread pain as defined by the criteria of the 1990 ACR (i.e. fibromyalgia)
* A lifetime history of spinal traumata (e.g. whiplash), surgery (e.g. laminectomy) or deformations (e.g. scoliosis)
* A lifetime history of respiratory, metabolic, neurologic, cardiovascular, inflammatory, orthopedic or rheumatologic diseases
* Concomitant therapies (i.e. rehabilitation, alternative medicine or therapies)
* Contra-indications for MRI (e.g. suffering from claustrophobia, the presence of metallic foreign material in the body, BMI >30kg/m²)
* Professional athletes
* Pregnant women
* Breastfeeding women
* Women given birth in the last year before enrolment

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Brain macro-structure | Baseline
  Whole brain T1-weighted structural MRI will be acquired.
Brain macro-structure | After low-load training phase (i.e. after 9th supervised treatment session) assessed at approximately 8 weeks
  Whole brain T1-weighted structural MRI will be acquired.
Brain macro-structure | After high-load training phase (i.e. after 18th supervised treatment session) assessed at approximately 13 weeks
  Whole brain T1-weighted structural MRI will be acquired.
Brain macro-structure | At 3 months follow-up
  Whole brain T1-weighted structural MRI will be acquired.
Brain micro-structure | Baseline
  Whole-brain T2-weighted images will be obtained.
Brain micro-structure | After low-load training phase (i.e. after 9th supervised treatment session) assessed at approximately 8 weeks
  Whole-brain T2-weighted images will be obtained.
Brain micro-structure | After high-load training phase (i.e. after 18th supervised treatment session) assessed at approximately 13 weeks
  Whole-brain T2-weighted images will be obtained.
Brain micro-structure | At 3 months follow-up
  Whole-brain T2-weighted images will be obtained.

SECONDARY OUTCOMES:
Functional brain connectivity | Baseline
  Resting-state functional MRI will be performed to acquire insight into subnetworks relating to sensorimotor control and pain processing.
Functional brain connectivity | After low-load training phase (i.e. after 9th supervised treatment session) assessed at approximately 8 weeks
  Resting-state functional MRI will be performed to acquire insight into subnetworks relating to sensorimotor control and pain processing.
Functional brain connectivity | After high-load training phase (i.e. after 18th supervised treatment session) assessed at approximately 13 weeks
  Resting-state functional MRI will be performed to acquire insight into subnetworks relating to sensorimotor control and pain processing.
Functional brain connectivity | At 3 months follow-up
  Resting-state functional MRI will be performed to acquire insight into subnetworks relating to sensorimotor control and pain processing.
Lumbar muscle structure | Baseline
  T1-weighted Dixon MRI will be performed.
Lumbar muscle structure | After low-load training phase (i.e. after 9th supervised treatment session) assessed at approximately 8 weeks
  T1-weighted Dixon MRI will be performed.
Lumbar muscle structure | After high-load training phase (i.e. after 18th supervised treatment session) assessed at approximately 13 weeks
  T1-weighted Dixon MRI will be performed.
Lumbar muscle structure | At 3 months follow-up
  T1-weighted Dixon MRI will be performed.
Lumbar muscle function | Baseline
  T2-weighted mf-MRI will be conducted.
Lumbar muscle function | After low-load training phase (i.e. after 9th supervised treatment session) assessed at approximately 8 weeks
  T2-weighted mf-MRI will be conducted.
Lumbar muscle function | After high-load training phase (i.e. after 18th supervised treatment session) assessed at approximately 13 weeks
  T2-weighted mf-MRI will be conducted.
Lumbar muscle function | At 3 months follow-up.
  T2-weighted mf-MRI will be conducted.
Lumbopelvic control | Baseline
  Lumbopelvic control will be examined by means of a clinical thoracolumbar dissociation test which assesses the quality of performance of lumbopelvic motion with limited motion at the thoracolumbar junction.
Lumbopelvic control | After low-load training phase (i.e. after 9th supervised treatment session) assessed at approximately 8 weeks
  Lumbopelvic control will be examined by means of a clinical thoracolumbar dissociation test which assesses the quality of performance of lumbopelvic motion with limited motion at the thoracolumbar junction.
Lumbopelvic control | After high-load training phase (i.e. after 18th supervised treatment session) assessed at approximately 13 weeks
  Lumbopelvic control will be examined by means of a clinical thoracolumbar dissociation test which assesses the quality of performance of lumbopelvic motion with limited motion at the thoracolumbar junction.
Lumbopelvic control | At 3 months follow-up.
  Lumbopelvic control will be examined by means of a clinical thoracolumbar dissociation test which assesses the quality of performance of lumbopelvic motion with limited motion at the thoracolumbar junction.
Lumbopelvic proprioception | Baseline
  To evaluate lumbar proprioception, the position-reposition accuracy of the lumbar spine will be determined.
Lumbopelvic proprioception | After low-load training phase (i.e. after 9th supervised treatment session) assessed at approximately 8 weeks
  To evaluate lumbar proprioception, the position-reposition accuracy of the lumbar spine will be determined.
Lumbopelvic proprioception | After high-load training phase (i.e. after 18th supervised treatment session) assessed at approximately 13 weeks
  To evaluate lumbar proprioception, the position-reposition accuracy of the lumbar spine will be determined.
Lumbopelvic proprioception | At 3 months follow-up.
  To evaluate lumbar proprioception, the position-reposition accuracy of the lumbar spine will be determined.
Anticipatory postural adjustments | Baseline
  To examine anticipatory postural adjustments (APAs) trunk muscle onset latencies in response to internal-induced perturbations will be measured by means of surface electromyography (EMG). APAs will be measured by inducing internal perturbations in the trunk muscles during a reliable and valid unilateral rapid arm movement task (RAM).
Anticipatory postural adjustments | After low-load training phase (i.e. after 9th supervised treatment session) assessed at approximately 8 weeks
  To examine anticipatory postural adjustments (APAs) trunk muscle onset latencies in response to internal-induced perturbations will be measured by means of surface electromyography (EMG). APAs will be measured by inducing internal perturbations in the trunk muscles during a reliable and valid unilateral rapid arm movement task (RAM).
Anticipatory postural adjustments | After high-load training phase (i.e. after 18th supervised treatment session) assessed at approximately 13 weeks
  To examine anticipatory postural adjustments (APAs) trunk muscle onset latencies in response to internal-induced perturbations will be measured by means of surface electromyography (EMG). APAs will be measured by inducing internal perturbations in the trunk muscles during a reliable and valid unilateral rapid arm movement task (RAM).
Anticipatory postural adjustments | At 3 months follow-up
  To examine anticipatory postural adjustments (APAs) trunk muscle onset latencies in response to internal-induced perturbations will be measured by means of surface electromyography (EMG). APAs will be measured by inducing internal perturbations in the trunk muscles during a reliable and valid unilateral rapid arm movement task (RAM).
Compensatory postural adjustments | Baseline
  To examine compensatory postural adjustments (CPAs), trunk muscle onset latencies in response to external-induced perturbations will be measured by means of surface electromyography (EMG). CPAs will be measured by using external perturbations of trunk muscles during a quick-force-release test (QFRT).
Compensatory postural adjustments | After low-load training phase (i.e. after 9th supervised treatment session) assessed at approximately 8 weeks
  To examine compensatory postural adjustments (CPAs), trunk muscle onset latencies in response to external-induced perturbations will be measured by means of surface electromyography (EMG). CPAs will be measured by using external perturbations of trunk muscles during a quick-force-release test (QFRT).
Compensatory postural adjustments | After high-load training phase (i.e. after 18th supervised treatment session) assessed at approximately 13 weeks
  To examine compensatory postural adjustments (CPAs), trunk muscle onset latencies in response to external-induced perturbations will be measured by means of surface electromyography (EMG). CPAs will be measured by using external perturbations of trunk muscles during a quick-force-release test (QFRT).
Compensatory postural adjustments | At 3 months follow-up
  To examine compensatory postural adjustments (CPAs), trunk muscle onset latencies in response to external-induced perturbations will be measured by means of surface electromyography (EMG). CPAs will be measured by using external perturbations of trunk muscles during a quick-force-release test (QFRT).
Nociceptive flexion reflex - threshold | Baseline
  The NFR will be elicited in the dominant leg by transcutaneous electrical stimulation of the sural nerve in its retromalleolar path using a stimulation bar electrode connected to a constant current stimulator. Surface EMG electrodes will be placed on the skin of the muscle belly of the ipsilateral biceps femoris.
Nociceptive flexion reflex - threshold | After low-load training phase (i.e. after 9th supervised treatment session) assessed at approximately 8 weeks
  The NFR will be elicited in the dominant leg by transcutaneous electrical stimulation of the sural nerve in its retromalleolar path using a stimulation bar electrode connected to a constant current stimulator. Surface EMG electrodes will be placed on the skin of the muscle belly of the ipsilateral biceps femoris.
Nociceptive flexion reflex - threshold | After high-load training phase (i.e. after 18th supervised treatment session) assessed at approximately 13 weeks
  The NFR will be elicited in the dominant leg by transcutaneous electrical stimulation of the sural nerve in its retromalleolar path using a stimulation bar electrode connected to a constant current stimulator. Surface EMG electrodes will be placed on the skin of the muscle belly of the ipsilateral biceps femoris.
Nociceptive flexion reflex - threshold | At 3 months follow-up
  The NFR will be elicited in the dominant leg by transcutaneous electrical stimulation of the sural nerve in its retromalleolar path using a stimulation bar electrode connected to a constant current stimulator. Surface EMG electrodes will be placed on the skin of the muscle belly of the ipsilateral biceps femoris.
Nociceptive flexion reflex - temporal summation | Baseline
  Five 1ms rectangular wave pulse train will be administered 3 times at a frequency of 2 Hz at a constant stimulation intensity. This procedure will be repeated 5 times.
Nociceptive flexion reflex - temporal summation | After low-load training phase (i.e. after 9th supervised treatment session) assessed at approximately 8 weeks
  Five 1ms rectangular wave pulse train will be administered 3 times at a frequency of 2 Hz at a constant stimulation intensity. This procedure will be repeated 5 times.
Nociceptive flexion reflex - temporal summation | After high-load training phase (i.e. after 18th supervised treatment session) assessed at approximately 13 weeks
  Five 1ms rectangular wave pulse train will be administered 3 times at a frequency of 2 Hz at a constant stimulation intensity. This procedure will be repeated 5 times.
Nociceptive flexion reflex - temporal summation | At 3 months follow-up
  Five 1ms rectangular wave pulse train will be administered 3 times at a frequency of 2 Hz at a constant stimulation intensity. This procedure will be repeated 5 times.
Conditioned pain modulation | Baseline
  The conditioning stimulus will comprise of immersion of the non-dominant hand until the proximal wrist crease in a hot circulating water bath of 45.5°C during 6 minutes. The test stimulus will comprise of pressure pain threshold (PPT) assessments (as described above) during and after completion of the conditioning stimulus. Before, after 2 min of immersion and 2 minutes after completion of immersion, the test stimulus will be repeated twice at each test location at the dominant body side.
Conditioned pain modulation | After low-load training phase (i.e. after 9th supervised treatment session) assessed at approximately 8 weeks
  The conditioning stimulus will comprise of immersion of the non-dominant hand until the proximal wrist crease in a hot circulating water bath of 45.5°C during 6 minutes. The test stimulus will comprise of pressure pain threshold (PPT) assessments (as described above) during and after completion of the conditioning stimulus. Before, after 2 min of immersion and 2 minutes after completion of immersion, the test stimulus will be repeated twice at each test location at the dominant body side.
Conditioned pain modulation | After high-load training phase (i.e. after 18th supervised treatment session) assessed at approximately 13 weeks
  The conditioning stimulus will comprise of immersion of the non-dominant hand until the proximal wrist crease in a hot circulating water bath of 45.5°C during 6 minutes. The test stimulus will comprise of pressure pain threshold (PPT) assessments (as described above) during and after completion of the conditioning stimulus. Before, after 2 min of immersion and 2 minutes after completion of immersion, the test stimulus will be repeated twice at each test location at the dominant body side.
Conditioned pain modulation | At 3 months follow-up
  The conditioning stimulus will comprise of immersion of the non-dominant hand until the proximal wrist crease in a hot circulating water bath of 45.5°C during 6 minutes. The test stimulus will comprise of pressure pain threshold (PPT) assessments (as described above) during and after completion of the conditioning stimulus. Before, after 2 min of immersion and 2 minutes after completion of immersion, the test stimulus will be repeated twice at each test location at the dominant body side.
Anxiety and depression | Baseline
  Hospital Anxiety and depression scale (HADS)
Anxiety and depression | After low-load training phase (i.e. after 9th supervised treatment session) assessed at approximately 8 weeks
  Hospital Anxiety and depression scale (HADS)
Anxiety and depression | After high-load training phase (i.e. after 18th supervised treatment session) assessed at approximately 13 weeks
  Hospital Anxiety and depression scale (HADS)
Anxiety and depression | At 3 months follow-up
  Hospital Anxiety and depression scale (HADS)
Physical activity | Baseline
  International physical activity questionnaire - long form (IPAQ-LF)
Physical activity | After low-load training phase (i.e. after 9th supervised treatment session) assessed at approximately 8 weeks
  International physical activity questionnaire - long form (IPAQ-LF)
Physical activity | After high-load training phase (i.e. after 18th supervised treatment session) assessed at approximately 13 weeks
  International physical activity questionnaire - long form (IPAQ-LF)
Physical activity | At 3 months follow-up.
  International physical activity questionnaire - long form (IPAQ-LF)
Pain coping | Baseline
  Pain coping inventory (PCI), Pain Catastrophizing Scale (PCS)
Pain coping | After low-load training phase (i.e. after 9th supervised treatment session) assessed at approximately 8 weeks
  Pain coping inventory (PCI), Pain Catastrophizing Scale (PCS)
Pain coping | After high-load training phase (i.e. after 18th supervised treatment session) assessed at approximately 13 weeks
  Pain coping inventory (PCI), Pain Catastrophizing Scale (PCS)
Pain coping | At 3 months follow-up
  Pain coping inventory (PCI), Pain Catastrophizing Scale (PCS)
Pain catastrophizing | Baseline
  Pain Catastrophizing Scale (PCS)
Pain catastrophizing | After low-load training phase (i.e. after 9th supervised treatment session) assessed at approximately 8 weeks
  Pain Catastrophizing Scale (PCS)
Pain catastrophizing | After high-load training phase (i.e. after 18th supervised treatment session) assessed at approximately 13 weeks
  Pain Catastrophizing Scale (PCS)
Pain catastrophizing | At 3 months follow-up
  Pain Catastrophizing Scale (PCS)
Pain vigilance and awareness | Baseline
  Pain vigilance and awareness questionnaire (PVAQ)
Pain vigilance and awareness | After low-load training phase (i.e. after 9th supervised treatment session) assessed at approximately 8 weeks
  Pain vigilance and awareness questionnaire (PVAQ)
Pain vigilance and awareness | After high-load training phase (i.e. after 18th supervised treatment session) assessed at approximately 13 weeks
  Pain vigilance and awareness questionnaire (PVAQ)
Pain vigilance and awareness | At 3 months follow-up
  Pain vigilance and awareness questionnaire (PVAQ)
Kinesiophobia | Baseline
  Tampa Scale for Kinesiophobia (TSK)
Kinesiophobia | After low-load training phase (i.e. after 9th supervised treatment session) assessed at approximately 8 weeks
  Tampa Scale for Kinesiophobia (TSK)
Kinesiophobia | After high-load training phase (i.e. after 18th supervised treatment session) assessed at approximately 13 weeks
  Tampa Scale for Kinesiophobia (TSK)
Kinesiophobia | At 3 months follow-up
  Tampa Scale for Kinesiophobia (TSK)
Health status | Baseline
  Short Form Health Survey-36 items (SF-36)
Health status | After low-load training phase (i.e. after 9th supervised treatment session) assessed at approximately 8 weeks
  Short Form Health Survey-36 items (SF-36)
Health status | After high-load training phase (i.e. after 18th supervised treatment session) assessed at approximately 13 weeks
  Short Form Health Survey-36 items (SF-36)
Health status | At 3 months follow-up
  Short Form Health Survey-36 items (SF-36)
Low back pain related pain | Baseline
  LBP related pain intensity will be evaluated by using an 11 point NRS
Low back pain related pain | After low-load training phase (i.e. after 9th supervised treatment session) assessed at approximately 8 weeks
  LBP related pain intensity will be evaluated by using an 11 point NRS
Low back pain related pain | After high-load training phase (i.e. after 18th supervised treatment session) assessed at approximately 13 weeks
  LBP related pain intensity will be evaluated by using an 11 point NRS
Low back pain related pain | At 3 months follow-up
  LBP related pain intensity will be evaluated by using an 11 point NRS
Low back pain related disability | Baseline
  The Roland Morris Disability Questionnaire will be used to evaluate disability.
Low back pain related disability | After low-load training phase (i.e. after 9th supervised treatment session) assessed at approximately 8 weeks
  The Roland Morris Disability Questionnaire will be used to evaluate disability.
Low back pain related disability | After high-load training phase (i.e. after 18th supervised treatment session) assessed at approximately 13 weeks
  The Roland Morris Disability Questionnaire will be used to evaluate disability.
Low back pain related disability | At 3 months follow-up
  The Roland Morris Disability Questionnaire will be used to evaluate disability.
Low back pain recurrence | At 6 months follow-up
  Self-report via telephone interview: (1) the number of episode(s), (2) the duration of the LBP episode(s), (3) pain intensity, measured with three NRS for average-, worst- and current pain during the LBP episode(s), (4) location and quality of pain (i.e. sharp, burning, etc. sensation), (5) subjects opinion about what caused the new episode of LBP, (6) degree of impairments in daily life activities due to the LBP, (7) whether participants sought treatment (i.e. physiotherapist, general practitioner, etc.) and (8) strategies to cope with the new LBP episode.
Low back pain recurrence | At 12 months follow-up
  Self-report via telephone interview: (1) the number of episode(s), (2) the duration of the LBP episode(s), (3) pain intensity, measured with three NRS for average-, worst- and current pain during the LBP episode(s), (4) location and quality of pain (i.e. sharp, burning, etc. sensation), (5) subjects opinion about what caused the new episode of LBP, (6) degree of impairments in daily life activities due to the LBP, (7) whether participants sought treatment (i.e. physiotherapist, general practitioner, etc.) and (8) strategies to cope with the new LBP episode.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica van Oosterwijck, Prof, Study Director — Ghent University, Pain in Motion
Locations (1):
- Ghent University, vakgroep revalidatiewetenschappen, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hartvigsen J, Hancock MJ, Kongsted A, Louw Q, Ferreira ML, Genevay S, Hoy D, Karppinen J, Pransky G, Sieper J, Smeets RJ, Underwood M; Lancet Low Back Pain Series Working Group. What low back pain is and why we need to pay attention. Lancet. 2018 Jun 9;391(10137):2356-2367. doi: 10.1016/S0140-6736(18)30480-X. Epub 2018 Mar 21. PMID 29573870
- [Background] Hurwitz EL, Randhawa K, Yu H, Cote P, Haldeman S. The Global Spine Care Initiative: a summary of the global burden of low back and neck pain studies. Eur Spine J. 2018 Sep;27(Suppl 6):796-801. doi: 10.1007/s00586-017-5432-9. Epub 2018 Feb 26. PMID 29480409
- [Background] Deyo RA. Diagnostic evaluation of LBP: reaching a specific diagnosis is often impossible. Arch Intern Med. 2002 Jul 8;162(13):1444-7; discussion 1447-8. doi: 10.1001/archinte.162.13.1444. No abstract available. PMID 12090877
- [Background] Iizuka Y, Iizuka H, Mieda T, Tsunoda D, Sasaki T, Tajika T, Yamamoto A, Takagishi K. Prevalence of Chronic Nonspecific Low Back Pain and Its Associated Factors among Middle-Aged and Elderly People: An Analysis Based on Data from a Musculoskeletal Examination in Japan. Asian Spine J. 2017 Dec;11(6):989-997. doi: 10.4184/asj.2017.11.6.989. Epub 2017 Dec 7. PMID 29279756
- [Background] Itz CJ, Geurts JW, van Kleef M, Nelemans P. Clinical course of non-specific low back pain: a systematic review of prospective cohort studies set in primary care. Eur J Pain. 2013 Jan;17(1):5-15. doi: 10.1002/j.1532-2149.2012.00170.x. Epub 2012 May 28. PMID 22641374
- [Background] da C Menezes Costa L, Maher CG, Hancock MJ, McAuley JH, Herbert RD, Costa LO. The prognosis of acute and persistent low-back pain: a meta-analysis. CMAJ. 2012 Aug 7;184(11):E613-24. doi: 10.1503/cmaj.111271. Epub 2012 May 14. PMID 22586331
- [Background] da Silva T, Mills K, Brown BT, Herbert RD, Maher CG, Hancock MJ. Risk of Recurrence of Low Back Pain: A Systematic Review. J Orthop Sports Phys Ther. 2017 May;47(5):305-313. doi: 10.2519/jospt.2017.7415. Epub 2017 Mar 29. PMID 28355981
- [Background] Goubert D, Meeus M, Willems T, De Pauw R, Coppieters I, Crombez G, Danneels L. The association between back muscle characteristics and pressure pain sensitivity in low back pain patients. Scand J Pain. 2018 Apr 25;18(2):281-293. doi: 10.1515/sjpain-2017-0142. PMID 29794309
- [Background] Ranger TA, Cicuttini FM, Jensen TS, Peiris WL, Hussain SM, Fairley J, Urquhart DM. Are the size and composition of the paraspinal muscles associated with low back pain? A systematic review. Spine J. 2017 Nov;17(11):1729-1748. doi: 10.1016/j.spinee.2017.07.002. Epub 2017 Jul 26. PMID 28756299
- [Background] Kregel J, Meeus M, Malfliet A, Dolphens M, Danneels L, Nijs J, Cagnie B. Structural and functional brain abnormalities in chronic low back pain: A systematic review. Semin Arthritis Rheum. 2015 Oct;45(2):229-37. doi: 10.1016/j.semarthrit.2015.05.002. Epub 2015 May 16. PMID 26092329
- [Background] Coppieters I, Meeus M, Kregel J, Caeyenberghs K, De Pauw R, Goubert D, Cagnie B. Relations Between Brain Alterations and Clinical Pain Measures in Chronic Musculoskeletal Pain: A Systematic Review. J Pain. 2016 Sep;17(9):949-62. doi: 10.1016/j.jpain.2016.04.005. Epub 2016 Jun 3. PMID 27263992
- [Background] Yuan C, Shi H, Pan P, Dai Z, Zhong J, Ma H, Sheng L. Gray Matter Abnormalities Associated With Chronic Back Pain: A Meta-Analysis of Voxel-based Morphometric Studies. Clin J Pain. 2017 Nov;33(11):983-990. doi: 10.1097/AJP.0000000000000489. PMID 28234752
- [Background] Brumagne S, Diers M, Danneels L, Moseley GL, Hodges PW. Neuroplasticity of Sensorimotor Control in Low Back Pain. J Orthop Sports Phys Ther. 2019 Jun;49(6):402-414. doi: 10.2519/jospt.2019.8489. PMID 31151373
- [Background] Moseley GL, Flor H. Targeting cortical representations in the treatment of chronic pain: a review. Neurorehabil Neural Repair. 2012 Jul-Aug;26(6):646-52. doi: 10.1177/1545968311433209. Epub 2012 Feb 13. PMID 22331213
- [Background] Kilgour AH, Todd OM, Starr JM. A systematic review of the evidence that brain structure is related to muscle structure and their relationship to brain and muscle function in humans over the lifecourse. BMC Geriatr. 2014 Jul 10;14:85. doi: 10.1186/1471-2318-14-85. PMID 25011478
- [Background] Goossens N, Rummens S, Janssens L, Caeyenberghs K, Brumagne S. Association Between Sensorimotor Impairments and Functional Brain Changes in Patients With Low Back Pain: A Critical Review. Am J Phys Med Rehabil. 2018 Mar;97(3):200-211. doi: 10.1097/PHM.0000000000000859. PMID 29112509
- [Background] Panjabi M, Abumi K, Duranceau J, Oxland T. Spinal stability and intersegmental muscle forces. A biomechanical model. Spine (Phila Pa 1976). 1989 Feb;14(2):194-200. doi: 10.1097/00007632-198902000-00008. PMID 2922640
- [Background] Panjabi MM. The stabilizing system of the spine. Part I. Function, dysfunction, adaptation, and enhancement. J Spinal Disord. 1992 Dec;5(4):383-9; discussion 397. doi: 10.1097/00002517-199212000-00001. PMID 1490034
- [Background] Panjabi MM. The stabilizing system of the spine. Part II. Neutral zone and instability hypothesis. J Spinal Disord. 1992 Dec;5(4):390-6; discussion 397. doi: 10.1097/00002517-199212000-00002. PMID 1490035
- [Background] Goubert D, Oosterwijck JV, Meeus M, Danneels L. Structural Changes of Lumbar Muscles in Non-specific Low Back Pain: A Systematic Review. Pain Physician. 2016 Sep-Oct;19(7):E985-E1000. PMID 27676689
- [Background] Danneels LA, Vanderstraeten GG, Cambier DC, Witvrouw EE, De Cuyper HJ. CT imaging of trunk muscles in chronic low back pain patients and healthy control subjects. Eur Spine J. 2000 Aug;9(4):266-72. doi: 10.1007/s005860000190. PMID 11261613
- [Background] D'hooge R, Cagnie B, Crombez G, Vanderstraeten G, Dolphens M, Danneels L. Increased intramuscular fatty infiltration without differences in lumbar muscle cross-sectional area during remission of unilateral recurrent low back pain. Man Ther. 2012 Dec;17(6):584-8. doi: 10.1016/j.math.2012.06.007. Epub 2012 Jul 10. PMID 22784801
- [Background] Cagnie B, Dhooge F, Schumacher C, De Meulemeester K, Petrovic M, van Oosterwijck J, Danneels L. Fiber Typing of the Erector Spinae and Multifidus Muscles in Healthy Controls and Back Pain Patients: A Systematic Literature Review. J Manipulative Physiol Ther. 2015 Nov-Dec;38(9):653-663. doi: 10.1016/j.jmpt.2015.10.004. Epub 2015 Nov 5. PMID 26547762
- [Background] Agten A, Stevens S, Verbrugghe J, Timmermans A, Vandenabeele F. Biopsy samples from the erector spinae of persons with nonspecific chronic low back pain display a decrease in glycolytic muscle fibers. Spine J. 2020 Feb;20(2):199-206. doi: 10.1016/j.spinee.2019.09.023. Epub 2019 Sep 27. PMID 31563580
- [Background] D'hooge R, Cagnie B, Crombez G, Vanderstraeten G, Achten E, Danneels L. Lumbar muscle dysfunction during remission of unilateral recurrent nonspecific low-back pain: evaluation with muscle functional MRI. Clin J Pain. 2013 Mar;29(3):187-94. doi: 10.1097/AJP.0b013e31824ed170. PMID 23369927
- [Background] Knox MF, Chipchase LS, Schabrun SM, Romero RJ, Marshall PWM. Anticipatory and compensatory postural adjustments in people with low back pain: a systematic review and meta-analysis. Spine J. 2018 Oct;18(10):1934-1949. doi: 10.1016/j.spinee.2018.06.008. Epub 2018 Jun 12. PMID 29906616
- [Background] Prins MR, Griffioen M, Veeger TTJ, Kiers H, Meijer OG, van der Wurff P, Bruijn SM, van Dieen JH. Evidence of splinting in low back pain? A systematic review of perturbation studies. Eur Spine J. 2018 Jan;27(1):40-59. doi: 10.1007/s00586-017-5287-0. Epub 2017 Sep 12. PMID 28900711
- [Background] D'hooge R, Hodges P, Tsao H, Hall L, Macdonald D, Danneels L. Altered trunk muscle coordination during rapid trunk flexion in people in remission of recurrent low back pain. J Electromyogr Kinesiol. 2013 Feb;23(1):173-81. doi: 10.1016/j.jelekin.2012.09.003. Epub 2012 Oct 15. PMID 23079004
- [Background] Geisser ME, Ranavaya M, Haig AJ, Roth RS, Zucker R, Ambroz C, Caruso M. A meta-analytic review of surface electromyography among persons with low back pain and normal, healthy controls. J Pain. 2005 Nov;6(11):711-26. doi: 10.1016/j.jpain.2005.06.008. PMID 16275595
- [Background] Hodges PW, Moseley GL. Pain and motor control of the lumbopelvic region: effect and possible mechanisms. J Electromyogr Kinesiol. 2003 Aug;13(4):361-70. doi: 10.1016/s1050-6411(03)00042-7. PMID 12832166
- [Background] Hodges PW. Core stability exercise in chronic low back pain. Orthop Clin North Am. 2003 Apr;34(2):245-54. doi: 10.1016/s0030-5898(03)00003-8. PMID 12914264
- [Background] Ebenbichler GR, Oddsson LI, Kollmitzer J, Erim Z. Sensory-motor control of the lower back: implications for rehabilitation. Med Sci Sports Exerc. 2001 Nov;33(11):1889-98. doi: 10.1097/00005768-200111000-00014. PMID 11689740
- [Background] Saragiotto BT, Maher CG, Yamato TP, Costa LO, Menezes Costa LC, Ostelo RW, Macedo LG. Motor control exercise for chronic non-specific low-back pain. Cochrane Database Syst Rev. 2016 Jan 8;2016(1):CD012004. doi: 10.1002/14651858.CD012004. PMID 26742533
- [Background] Macedo LG, Saragiotto BT, Yamato TP, Costa LO, Menezes Costa LC, Ostelo RW, Maher CG. Motor control exercise for acute non-specific low back pain. Cochrane Database Syst Rev. 2016 Feb 10;2(2):CD012085. doi: 10.1002/14651858.CD012085. PMID 26863390
- [Background] Foster NE, Anema JR, Cherkin D, Chou R, Cohen SP, Gross DP, Ferreira PH, Fritz JM, Koes BW, Peul W, Turner JA, Maher CG; Lancet Low Back Pain Series Working Group. Prevention and treatment of low back pain: evidence, challenges, and promising directions. Lancet. 2018 Jun 9;391(10137):2368-2383. doi: 10.1016/S0140-6736(18)30489-6. Epub 2018 Mar 21. PMID 29573872
- [Background] Tsao H, Druitt TR, Schollum TM, Hodges PW. Motor training of the lumbar paraspinal muscles induces immediate changes in motor coordination in patients with recurrent low back pain. J Pain. 2010 Nov;11(11):1120-8. doi: 10.1016/j.jpain.2010.02.004. PMID 20434958
- [Background] Liu KP, Chan CC, Lee TM, Hui-Chan CW. Mental imagery for promoting relearning for people after stroke: a randomized controlled trial. Arch Phys Med Rehabil. 2004 Sep;85(9):1403-8. doi: 10.1016/j.apmr.2003.12.035. PMID 15375808
- [Background] Tsao H, Galea MP, Hodges PW. Driving plasticity in the motor cortex in recurrent low back pain. Eur J Pain. 2010 Sep;14(8):832-9. doi: 10.1016/j.ejpain.2010.01.001. Epub 2010 Feb 23. PMID 20181504
- [Background] Masse-Alarie H, Beaulieu LD, Preuss R, Schneider C. Influence of paravertebral muscles training on brain plasticity and postural control in chronic low back pain. Scand J Pain. 2016 Jul;12:74-83. doi: 10.1016/j.sjpain.2016.03.005. Epub 2016 May 11. PMID 28850499
- [Background] Taubert M, Lohmann G, Margulies DS, Villringer A, Ragert P. Long-term effects of motor training on resting-state networks and underlying brain structure. Neuroimage. 2011 Aug 15;57(4):1492-8. doi: 10.1016/j.neuroimage.2011.05.078. Epub 2011 Jun 7. PMID 21672633
- [Background] Taubert M, Draganski B, Anwander A, Muller K, Horstmann A, Villringer A, Ragert P. Dynamic properties of human brain structure: learning-related changes in cortical areas and associated fiber connections. J Neurosci. 2010 Sep 1;30(35):11670-7. doi: 10.1523/JNEUROSCI.2567-10.2010. PMID 20810887
- [Background] Tavor I, Botvinik-Nezer R, Bernstein-Eliav M, Tsarfaty G, Assaf Y. Short-term plasticity following motor sequence learning revealed by diffusion magnetic resonance imaging. Hum Brain Mapp. 2020 Feb 1;41(2):442-452. doi: 10.1002/hbm.24814. Epub 2019 Oct 9. PMID 31596547
- [Background] Draganski B, Gaser C, Busch V, Schuierer G, Bogdahn U, May A. Neuroplasticity: changes in grey matter induced by training. Nature. 2004 Jan 22;427(6972):311-2. doi: 10.1038/427311a. No abstract available. PMID 14737157
- [Background] Boyke J, Driemeyer J, Gaser C, Buchel C, May A. Training-induced brain structure changes in the elderly. J Neurosci. 2008 Jul 9;28(28):7031-5. doi: 10.1523/JNEUROSCI.0742-08.2008. PMID 18614670
- [Background] Scholz J, Klein MC, Behrens TE, Johansen-Berg H. Training induces changes in white-matter architecture. Nat Neurosci. 2009 Nov;12(11):1370-1. doi: 10.1038/nn.2412. Epub 2009 Oct 11. PMID 19820707